CLINICAL TRIAL: NCT05332743
Title: A Multi-center, Single-arm Prospective Study to Evaluate the Safety and Efficacy of a Nutraceutical Supplement With Vegan Botanicals in Females With Self-Perceived Thinning Hair
Brief Title: Nutraceutical Supplement With Vegan Botanicals in Females With Self-Perceived Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NW-VW-01
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hair Thinning
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: 6-month, multi-center, single-arm prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutraceutical Dietary Supplement (Experimental): Nutraceutical Dietary Supplement capsules are comprised of primary and secondary ingredients, designed to restore hair health from the inside out. In addition to the necessary vitamins, minerals, proteins to support the nutritional needs of hair.
  Interventions: Dietary Supplement: Nutrafol Vegan Women's Hair Supplement

INTERVENTIONS:
Dietary Supplement: Nutrafol Vegan Women's Hair Supplement — Nutrafol's Vegan Women's Hair Supplement with patented Synergen Complex® is a blend of proprietary formulation of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant and DHT-inhibiting properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. These ingredients include Sensoril Ashwagandha, Curcumin, Saw Palmetto, 20% Tocotrienol/Tocopherol complex, and capsaicin in combination with other vegan nutrients used to support hair health such as Pea Sprout Extract, Bamboo, and a new innovative Maldavian Dragonhead flower extract.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of a vegan nutraceutical supplement with standardized botanicals in females leading a more plant-based lifestyle with self-perceived thinning hair

DETAILED DESCRIPTION:
Hair loss is a common condition affecting both men and women that is more recently understood to be the result of multiple causes. Although it is generally a benign condition, hair loss can have a significant, detrimental impact on self-esteem, psychosocial functioning and the overall quality of life of affected individuals. It can also represent a substantial financial burden on individuals seeking treatment.

This is a 6-month, multi-center, single-arm prospective interventional study in adult female subjects who follow a plant-based diet with self-perceived hair thinning as confirmed by a dermatologist. The objective of this study is to assess the efficacy and safety of novel women's vegan supplement for hair growth.

ELIGIBILITY:
Inclusion Criteria:

1. Females of all Fitzpatrick skin, and hair types between 18-50 years of age with self-perceived thinning, confirmed by a dermatologist.
2. Females leading a more plant-based lifestyle as of the last 3 months or longer according to the following categories: Vegetarian, Lacto-vegetarian, Ovo-Vegetarian, Lacto-ovo Vegetarian, Vegan, Raw Vegan, Pescatarian, Pollotarian, Flexitarian/Semi-Vegetarian
3. Willing and able to adhere to the same dietary lifestyles for the duration of the study
4. Able to understand and sign an informed consent agreement and photo release form approved by the Institutional Review Board
5. General good health, as determined by the Investigator or qualified sub-investigator
6. Willing and able to attend all study visits and comply with the test product daily instructions.
7. Willing to maintain the same hair length, hairstyle, and coloring practices for the duration of the study. Subjects who have color-treated hair must have the color treatment performed at the same time interval prior to each visit.
8. Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth).
9. Willing and able to cooperate with the requirements of the study.
10. Able to complete and understand the various rating instruments.

Exclusion Criteria:

1. Individuals who are pregnant, planning a pregnancy, nursing, or within 1-year post-partum.
2. Individuals who have experienced serious complications due to COVID-19 previously or during the study as determined by the investigator.
3. Clinical diagnosis of hair loss disorder such as alopecia areata, or scarring forms of alopecia.
4. Individuals who have had a history of any acute or chronic disease that could interfere with or increase the risk on study participation
5. Individuals who have had a history of any acute or chronic medical or hair condition that could affect study results, such as a history of disordered eating
6. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
7. Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), infection, cuts, and/ or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator or qualified sub-investigator, might put the subject at risk or interfere with the study conduct or evaluations.
8. History of surgical correction of hair loss on the scalp (i.e., hair transplant).
9. Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 6 months prior to the Baseline Visit.
10. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study (the initiation of HRT or birth control should not have been associated with the initiation of hair loss/thinning).
11. History of burning, flaking, itching, and stinging of the scalp.
12. History of malignancy (except cutaneous squamous cell carcinoma and basal cell carcinoma) or currently undergoing chemotherapy or radiation treatments.
13. A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that in the opinion of the Investigator or qualified sub-investigator may interfere with the study treatment.
14. A known history of unstable or chronic depression or bipolar disease or any other condition that may impact the subject's participation in the opinion of the investigator or qualified sub-investigator.
15. A known allergy to any of the ingredients in the investigational product.
16. Utilization of low-level lasers for hair growth in the last three months.
17. Any condition that the Investigator thinks may put the subject at risk or interfere with their participation in the study or study results.
18. Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day.
19. Use of any medications or medicated shampoos that are known to potentially cause hair loss or affect hair growth, as determined by the Investigator or qualified sub-investigator.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Change in terminal hair counts at Day 180 relative to baseline (Day 0) | 180 Days
  Terminal Hair Counts

SECONDARY OUTCOMES:
Change in total, terminal and vellus and hair counts compared to baseline (Day 0) | 180 Days
  All Hair Counts
Change in Investigator Hair Quality Global Improvement Scale & Investigator Hair Growth Global Improvement Scale assessed by physician using standardized 2-D photographs compared to baseline. | 180 Days
  Investigator Score using a 0 to 10 VAS scale
Hair shedding pull test compared to baseline. | 180 Days
  Hair Pull Test
Subjective assessments of change in hair growth, appearance, and satisfaction measured with Subject Quality of Life Assessment | 180 Days
  Subject self-assessments of satisfaction and perception using a 4-pt scale
Compiled side effects, including all expected or unexpected side effects | All visits until 180 Days
  All side effects occurring during the study, categorized by severity (Mild, moderate, severe) and relatedness to the study product or participation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Integrative Skin Science and Research, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sivamani RK, Ablon G, Nong Y, Maloh J, Hazan A, Raymond I. A Prospective, Multi-Center Study to Evaluate the Safety and Efficacy of a Vegan Nutraceutical to Improve Hair Growth and Quality in Females Following a Plant-Based Diet. J Drugs Dermatol. 2024 Aug 1;23(8):661-668. doi: 10.36849/JDD.8421. PMID 39093662